CLINICAL TRIAL: NCT05863182
Title: JUNTOS (TOGETHER): Development of a Family-based Latino Youth Use Preventive Intervention
Brief Title: JUNTOS Familia Preventive Intervention
Acronym: Juntos
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00000702-MOD03
Record Dates: First submitted 2023-04-07; First posted 2023-05-17 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Alcohol Use, Underage
Keywords: Family; Latino; alcohol use; prevention; racism
MeSH Terms: conditions — Underage Drinking; Alcohol Drinking; Racism

STUDY DESIGN:
Intervention Model Description: cluster rct - will randomly assign 1/5 schools to serve as intervention school and 1/5 schools to serve as control school.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Students and parents attending the intervention school, will participate in the family-based intervention.
  Interventions: Behavioral: Juntos Familia Family based intervention
- Comparison Group (No Intervention): Students and parents attending the non-intervention school will not receive the intervention and serve as comparison group.

INTERVENTIONS:
Behavioral: Juntos Familia Family based intervention — Students and parents will participate in weekly 2.5 hour sessions around topics related to managing experiences with prejudice, discrimination and racism.
  Arms: Intervention Group

SUMMARY:
The primary objective of this study is to develop and pilot-test a family-based Latino youth alcohol use preventive intervention for Latino youth (ages 14-16) and one of their parents. The preventive intervention will equip youth, parents, and families with skills to manage stress related to prejudice, discrimination, and racism as a means to reduce Latino youth alcohol use risk. Informed by ecodevelopmental, social norms, family stress, stress and coping theories, and racial socialization theories, the central hypothesis is that active coping skills can buffer against the negative effect of social stressors (i.e., experiences related to prejudice, discrimination, and racism) on youth alcohol outcomes/related risks/cognitions; and active coping skills can offset the negative effect of social stress on parental adjustment, family functioning and parenting behaviors, thereby reducing youth alcohol use risk. Using an iterative approach to intervention development, within a mixed-method research design, the purpose of this study is to construct intervention sessions that impart active coping skills to better manage social stress related to prejudice, discrimination, and racism. In Aim 1, we will use qualitative methods to inform the development of intervention sessions that target coping with prejudice, discrimination, and racism. I will conduct focus groups with youth (5 groups, n=6-8) and parents (5 groups, n=6-8) to identify how youth and parents experience and cope with perceived ethnic discrimination; the skills and resources they would like to further develop; and to seek input regarding the structure and logistics of the intervention. In Aim 2, we will create a family-based youth alcohol use preventive intervention curriculum that targets coping with prejudice, discrimination, and racism. I will identify strategies used in existing preventive interventions and draw from Aim 1 qualitative findings to develop tentative intervention sessions. We will then conduct focus groups with youth (5 groups, n=6-8) and parents (5 groups, n=6-8) to seek feedback on tentative intervention sessions. We will then integrate focus group data into the intervention curriculum and modify it accordingly and develop manuals in English and Spanish. In Aim 3, we will pilot test the intervention among Latino families (i.e., one youth and one parent) in Texas. We will pilot test the intervention with 60 families (i.e., youth-parent dyads; N=30 intervention group; N = 30 comparison group) from high schools in the Austin Independent School District to a) assess intervention feasibility and acceptability, and b) determine preliminary effect size estimates for the intervention's promise to improve youth and parent coping skills, family functioning, parenting behaviors, and youth alcohol outcomes.

DETAILED DESCRIPTION:
SCHOOL SELECTION FOR QUASI-EXPERIMENTAL GROUP DESIGN. For aim 4, we have selected two out of five high schools that are closely are closely matched on the following criteria: 1) % Latino student enrollment (85.6 and 84.7), 2) % of students classified as economically disadvantaged (83 and 87), 3) Student achievement scores (66 and 69), 4) Student attendance scores (92 and 93), and 5) Student mobility rate (25.8 and 25.1). The matching of the two pilot study schools on these criteria, will allow us to eliminate any potential confounds that might preclude us from teasing apart the effects of the intervention from potential confounding school level effects. If the proposed intervention shows promise, we will be able to systematically test for school level effects in a larger, future study. We then propose to randomly assign one of the two schools to serve as intervention school and one of the two schools to serve as comparison school. The random assignment of one school to serve as intervention and one school to serve as comparison school will demonstrate the feasibility of randomization for a future larger study and will eliminate concerns about crossover and contamination.

Families from the intervention school (N = 30) will then be assigned to one of three intervention groups, each consisting of about 10 families (i.e., one youth and one parent), based on their language preference (English vs. Spanish). These families will then participate in the 9 week pilot intervention and fill-out a pre- and post-assessment battery.

Families from the comparison school (N = 30) will receive weekly information packages and fill out the pre- and post-assessment battery in the same week as the intervention school families.

For both groups, we will aim towards equal representation of boys and girls as well as U.S. and foreign-born youth. In line with the academic calendar of all the schools, we will aim to deliver the intervention from January to May to avoid delays due to school holidays and vacation.

Intervention Families will receive intervention sessions designed in PHASES 1-3. Sessions will be delivered in English or Spanish, based on participants' language preferences. We will conduct three groups (10 families and 2 facilitators/group). Although the time and location will be determined after study PHASE 3, based on my discussions with AISD, intervention sessions may be offered after school in a safe room. Incentives will include weekly non-monetary incentives, starting with small incentives (e.g., pens) and increasing the incentive value in later weeks (e.g., t-shirts). Each session will include a meal. Also, the time and location of the intervention will be determined based on the qualitative interview feedback. Participants will receive $30 for each completed assessment. Intervention session content will be delivered through short presentations, small/large group discussions, role-plays, exercises and practice of new skills. Each session will include home practice of new skills. Sessions will be digitally recorded. Recording will be used for future intervention refinement. Participants will be asked to respect the privacy of other group members. Facilitators: The PI will lead intervention sessions with a bilingual facilitator. The PI will, in consultation with co-primary mentors, Martinez and Marsiglia, train the facilitator by reviewing the intervention manual, emphasizing the purpose of each intervention component session and the need to not modify the manual. We will conduct mock intervention sessions and provide in-person feedback.

Comparison Families will receive 8 to 10 weekly information packages about the college application process. An information package may provide information about the application timeline and planning process. Participants will receive the information packages the same week the intervention families meet and sign a receipt for each package. Incentives: Comparison families will receive the same incentives as intervention families: weekly non-monetary incentives for picking up information packages and $30 for each completed assessment.

.2.

STATISTICAL DESIGN & POWER CONSIDERATIONS.

We will evaluate the feasibility and acceptability of the intervention with the following measures: number of families screened and enrolled per week, retention rates of intervention and comparison families, duration of assessment surveys and missing data, proportion of families who complete protocols for intervention and comparison intervention families, attendance at intervention sessions, preferred language for the intervention and comparison families, intervention engagement and interest, and reports of perceived barriers and facilitators for intervention participation.

We will also estimate whether the intervention shows promise on improving youth and parent coping skills, family functioning, and parenting behaviors and whether it shows promise in preventing youth alcohol outcomes and cognitions. The primary outcome of interest is coping skills. We will estimate the effect of the intervention on coping skills separately for youth and parents. Secondary outcomes include family functioning, parenting behaviors, alcohol use/related risks and alcohol related cognitions. We will estimate the effect of the intervention on family functioning, parenting behaviors, alcohol use/related risk and alcohol related cognitions separately for youth and parents.

In all intervention impact analyses, student and family outcomes will be compared for the intervention and comparison groups using an intention to treat (ITT) approach. We will use a generalized linear modeling framework, where post-intervention outcome measures will be regressed on an indicator variable for intervention versus comparison group status, while statistically controlling for baseline levels of coping skills, ethnic discrimination, and demographic variables.

Intervention impact estimates will be translated into standardized effect size indices (e.g., standardized mean differences, risk ratios) to facilitate interpretation of the magnitude and direction of potential intervention effects. Multiplicative interaction terms will be added to the generalized linear models to explore possible differential effects of the intervention on coping skills, family functioning, parenting behaviors, and alcohol outcomes and cognitions based on dosage and demographic variables.

Missing data will be handled with multiple imputation or full-information maximum likelihood-based approaches, presuming the data can be reasonably assumed to be missing at random. Should missing data or attrition be associated with covariates, appropriate covariates will be included in all impact analyses.

Given the exploratory nature of the proposed study, the moderate sample size, and a desire to detect early signs of promise of the intervention, we will focus on effect size estimates (e.g., 95% confidence intervals, standardized mean differences, Cohen's f), rather than on statistical significance. Co-primary mentor Martinez was able to identify beneficial effects of Nuestras Familias on parenting and youth outcomes with a sample of 73 families and such we believe that our sample size of 60 families will allow us to detect signs of promise of the intervention. Focusing on effect size estimates in this pilot feasibility study will allow me to plan a formal test of the intervention in a randomized trial (R01) to assess the efficacy of the intervention, isolate school level effects on intervention outcomes, and examine mediating and moderating mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* adolescents and caregivers (i.e., parents) in all of the study phases.
* adolescents between the ages 14 and 16, enrolled in 9th or 10th grade.
* adolescents must identify as "Hispanic," "Latino," or pan-ethnic labels.
* caregivers/parents with a 9th or 10th grade adolescent living at home.

B. SAMPLING/SCHOOL SELECTION.

* Austin Independent School District (AISD) for this project.
* Five high schools who meet the inclusion criteria:

  1. a high proportion of Latino students (>70%).
  2. a high proportion of students classified as economically disadvantaged (>50%).
  3. school enrollment of at least 1000 student.

Exclusion Criteria:

* Non Hispanic students and parents;
* Any Hispanic students and parents who don't meet above criteria.

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2024-08-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Coping Skills (Pre-assessment; week 1) | Pre-assessment (week 1)
  COPING SKILLS will be assessed via the COPE, a multidimensional assessment of active and avoidant coping strategies. Youth and parents report the frequency of using a given coping strategy: 1 (Not at All) to 4 (A Lot). We will assess discrimination specific active and avoidant coping with the Coping with Discrimination Scale. The CDS is a modified version of the COPE and includes 18 items assessing general and 7 items assessing discrimination specific coping strategies. We will also use the General Help-Seeking Questionnaire (GHSQ), which taps into youth and parents' social support seeking. The GHSQ provides participants with a list of people from whom parents and youth seek help. Participants rate on a scale from 1 (Extremely Unlikely) to 7 (Extremely Likely) their likelihood of seeking help. Lastly, we will assess youth-parent communication with 6 items from the racial socialization scale. Participants rate on a scale 1 (Very Unlikely) to 5 (Very Likely) their racial socialization.
Coping Skills (Post-assessment; weeks 16-20) | Pre-assessment (weeks 16-20)
  COPING SKILLS will be assessed via the COPE, a multidimensional assessment of active and avoidant coping strategies. Youth and parents report the frequency of using a given coping strategy: 1 (Not at All) to 4 (A Lot). We will assess discrimination specific active and avoidant coping with the Coping with Discrimination Scale which is a modified version of the COPE and includes 18 items assessing general and 7 items assessing discrimination specific coping strategies. We will also use the General Help-Seeking Questionnaire (GHSQ), which taps into youth and parents' social support seeking. The GHSQ provides participants with a list of people from whom parents and youth seek help. Participants rate on a scale from 1 (Extremely Unlikely) to 7 (Extremely Likely) their likelihood of seeking help. Lastly, we will assess youth-parent communication with 6 items from the racial socialization scale. Participants rate on a scale 1 (Very Unlikely) to 5 (Very Likely) their racial socialization.

SECONDARY OUTCOMES:
Alcohol Use Outcomes (Pre-assessment; week 1) | Pre-assessment (week 1)
  Past-year alcohol consumption and alcohol-related problems will be assessed with 10 items from the Alcohol Use Disorder Identification Test (AUDIT). Two subscales from the Comprehensive International Diagnostic Interview Brief Form (CIDI-BF) will be used to assess for adolescents past-year alcohol abuse and alcohol dependence. Four adapted questions from the Monitoring the Future Survey (MTF) will assess adolescent self-reports of recent alcohol use in the 14, 30 days, and 90 days. Four adapted questions from the MTF will assess adolescents' reports of being drunk in the past 14 days, 30 days, and 90 days prior to assessment. Eight questions from the Youth Risk Behavior Surveillance Survey will ask adolescents about their past 14 day, 30 day, and 90 day frequency of drunk driving and riding with a drunk driver. Sixteen items from the Short-Rutgers Alcohol Program Index (S-RAPI) will assess the frequency of alcohol-related negative consequences.
Alcohol Use Outcomes (Post-assessment; week 16-20) | Post-assessment (week 16-20)
  Past-year alcohol consumption and alcohol-related problems will be assessed with 10 items from the Alcohol Use Disorder Identification Test (AUDIT). Two subscales from the Comprehensive International Diagnostic Interview Brief Form (CIDI-BF) will be used to assess for adolescents past-year alcohol abuse and alcohol dependence. Four adapted questions from the Monitoring the Future Survey (MTF) will assess adolescent self-reports of recent alcohol use in the 14, 30 days, and 90 days. Four adapted questions from the MTF will assess adolescents' reports of being drunk in the past 14 days, 30 days, and 90 days prior to assessment. Eight questions from the Youth Risk Behavior Surveillance Survey will ask adolescents about their past 14 day, 30 day, and 90 day frequency of drunk driving and riding with a drunk driver. Sixteen items from the Short-Rutgers Alcohol Program Index (S-RAPI) will assess the frequency of alcohol-related negative consequences.
Family Functioning and Parenting Behaviors (Pre-assessment; week 1) | Pre-assessment (week 1)
  Family cohesion will be measured with six items from the Family Relations Scale which taps into youth and parent perceptions of feeling close and connected with each other. We will assess adolescent-parent communication with 20 items from the family communication scale which ask parents and youth about the degree to which they communicate with each other. We will assess parent and youth perceptions of positive and involved parenting behaviors with the Parenting Practices scale. Six items from the Parental Ethnic-Racial Socialization Scale will assess parent-youth communication regarding discrimination and parents' tendency to prepare their youth to navigate prejudice, discrimination, and racism.
Family Functioning and Parenting Behaviors (Post-assessment; weeks 16-20) | Post-assessment (week 16-20)
  Family cohesion will be measured with six items from the Family Relations Scale which taps into youth and parent perceptions of feeling close and connected with each other. We will assess adolescent-parent communication with 20 items from the family communication scale which ask parents and youth about the degree to which they communicate with each other. We will assess parent and youth perceptions of positive and involved parenting behaviors with the Parenting Practices scale. Six items from the Parental Ethnic-Racial Socialization Scale will assess parent-youth communication regarding discrimination and parents' tendency to prepare their youth to navigate prejudice, discrimination, and racism.

IPD SHARING:
Plan to Share IPD: Undecided
To be determined once enrollment occurs.